CLINICAL TRIAL: NCT00372307
Title: Efficacy and Safety of Pimecrolimus for the Treatment of Vitiligo Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003/275
Record Dates: First submitted 2006-09-04; First posted 2006-09-06 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Vitiligo Vulgaris
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Application of pimecrolimus

SUMMARY:
Patients with vitiligo vulgaris are treated with Pimecrolimus twice a day during 6 months. After a baseline visit, patient returns for a control visit after 3 and 6 months of treatment. One reference lesion is clinically evaluated with pictures.

ELIGIBILITY:
Inclusion Criteria:

* Active or stable vitiligo vulgaris
* lesions at head or neck + maximum 10% lesions at the rest of the body

Exclusion Criteria:

* Topica during last 2 weeks
* Photo(chemo)therapy during last 4 weeks
* Segmentary vitiligo

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26
Dates: Start 2004-05; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Repigmentation percentage of the reference lesion after 6 months.

SECONDARY OUTCOMES:
Number of patients with repigmentation after 3 and 6 months.
Repigmentation percentage of the reference lesion after 3 months.
Adverse events (month 3 and 6).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Naeyaert, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Background] Boone B, Ongenae K, Van Geel N, Vernijns S, De Keyser S, Naeyaert JM. Topical pimecrolimus in the treatment of vitiligo. Eur J Dermatol. 2007 Jan-Feb;17(1):55-61. doi: 10.1684/ejd.2007.0093. Epub 2007 Feb 27. PMID 17324829
- See also: Website of the University Hospital Ghent — http://www.uzgent.be